CLINICAL TRIAL: NCT00594906
Title: Use of Teriparatide to Accelerate Fracture Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to poor enrollment.
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Edward Puzas, Dr., University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50AR054041 (NIH); P50AR054041 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2013-03

CONDITIONS: Pelvic Fracture
Keywords: Fracture Healing; Teriparatide; Forteo; Pelvic Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection (Active Comparator): 30 participants will receive teriparatide (Forteo) injection pens.
  Interventions: Drug: Teriparatide
- Placebo (Placebo Comparator): 30 participants will receive placebo injection pens.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
  Other Names: Forteo
  Arms: Injection
Drug: Placebo — Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of the drug teriparatide to the effect of placebo on pelvic fracture healing.

DETAILED DESCRIPTION:
Teriparatide is a man-made form of a naturally occurring hormone called parathyroid. It increases bone density and bone strength to help prevent fractures and can be used to treat osteoporosis in people who have a high risk of bone fracture. The purpose of this study is to compare the effect of teriparatide to the effect of placebo on pelvic fracture healing.

This study will last 16 weeks. Participants will be randomly assigned to receive either teriparatide or placebo for the duration of the study. Participants will also be given calcium and vitamin D supplements to take daily throughout the study. At 4-week intervals, participants will undergo functional evaluations that will include the instrumented sit-to-stand test, the timed-up-and-go, and a gait velocity test. Participants will also undergo a DXA scan upon enrollment; undergo a CT evaluation upon enrollment and 16 weeks post-fracture; and complete specific pain, self-perceived function, mental status, and depression scales throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Females must be menopausal (no menses within the last 12 months)
* Low energy fragility fractures of the pelvis, including anterior column, posterior column, inferior or superior rami, or sacrum
* Maximum of 2 weeks post fracture
* Mental status consistent with completing the study protocol

Exclusion Criteria:

* Currently receiving any treatment for osteoporosis, including estrogen and estrogenic-like compounds
* Received radiation treatment to any site at any time in the past
* Received chemotherapy for cancer at any time in the past
* Any active cancer
* Surgical repair (or attempted repair) of the fracture site in the pelvis
* Use of any bone-active medications
* Use of anticonvulsant therapy
* Use of immunosuppressants
* Any renal, gastrointestinal, liver, or metabolic bone disease
* Pregnancy
* High calcium, parathyroid hormone, or alkaline phosphatase, as based on laboratory results

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Edward Puzas, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Forteo Injection: 30 participants will receive teriparatide (Forteo) injection pens.
  Teriparatide : Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
- Placebo Injection: 30 participants will receive placebo injection pens.
  Placebo : Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
Period: Overall Study
Arm/Group | Forteo Injection | Placebo Injection
Started | 7 | 3
Completed | 6 | 1
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Injection: 30 participants will receive teriparatide (Forteo) injection pens.
  Teriparatide : Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
- Placebo: 30 participants will receive placebo injection pens.
  Placebo : Daily 20-mcg subcutaneous injections for the duration of the study (16 weeks)
- Total: Total of all reporting groups
Arm/Group | Injection | Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (14) | 66 (5) | 75 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Healing of a Fracture From a Low Energy Fall
Description: Callus formation at the fracture site as defined by a CT scan to determine healing (early/beginning callus formation) or healed (complete callus formation)
Time Frame: Measured at 16 weeks
Measure: Number; unit: participants
Groups:
- Placebo Patients: Patients who recieved Placebo injections.
- Forteo Patients: Patients who recieved Forteo Injections.
Arm/Group | Placebo Patients | Forteo Patients
Number analyzed (Participants) | 3 | 7
participants
  Healed | 0 | 1
  Healing | 1 | 4
  Did not compelte CT scan | 2 | 2

ADVERSE EVENTS:
Groups:
- Forteo Injection: Patients who randomized to the study drug, Forteo
- Placebo Injection: Patients who were randomized to Placebo
Arm/Group | Forteo Injection | Placebo Injection
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 1/7 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forteo Injection (N=7) | Placebo Injection (N=3)
Fall (General disorders) | 1 (1) | 0 (0) — Px hospitalized day after consent-fell on hip/head. Suffered 3rd cranial nerve infarction,discharged. Returned to ED complaining of both legs, increased confusion and UTI. Treated for all and discharged. Patient fell again, suffered head laceration.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes